CLINICAL TRIAL: NCT01459822
Title: MiRNAhs in the Evaluation of the Value of Sepsis Prognosis Dynamics Observational Research
Brief Title: MiRNAs Evaluate the Prognosis of Sepsis by Dynamic Study
Acronym: METPSDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Other Study IDs: 301PLAGH-20110824005
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-08

CONDITIONS: Sepsis
Keywords: sepsis; miRNA
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — human serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Survival Group
- Death Group

SUMMARY:
Sepsis is a common cause of death in intensive care unit, timely and accurate diagnosis and treatment directly affect the survival rate. MiRNA is a post-transcriptional small RNA which regulate mRNA expression. The present study was designed to observe the selected miRNA expression which evaluate the sepsis prognosis in the progression of sepsis in order to be a new target for the treatment of sepsis.

DETAILED DESCRIPTION:
The study is a non-intervention observational study. Purpose of this study is to observe some selected miRNA expression which evaluate the sepsis prognosis in the progression of sepsis . The investigators will collect serum samples from patients with sepsis in SICU, RICU and EICU on the 1st、3rd、5th、7th、10th、14th day of 301 Hospital since November 2011 , and then use mirVana PARIS kit extract total RNA and use qRT-PCR detect miRNAS expression in serum which can evaluate the prognosis of sepsis, and statistical analysis the miRNAS expression correlation with SOFA score.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of sepsis
* Patients who agree with the study

Exclusion Criteria:

* Aged <18 years;
* Into the group who died within 24 hours;
* Agranulocytosis (<0.5 × 109 / L);
* Combined HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: within 24 hours after admited in ICU
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-07 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | 28days after admited in ICU

CONTACTS AND LOCATIONS:
Overall Officials: LiXin Xie, doctor, Study Director — Pneumology Department of chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Haidian, China